CLINICAL TRIAL: NCT03226587
Title: Acute Effects of Whole Body Blue Light Exposure on Blood Pressure, Endothelial Function and Vascular Stiffness
Brief Title: Acute Effects of Whole Body Blue Light Exposure on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Philips GmbH, Innovative Technologies, Aachen (Unknown); Klinik für Unfall - und Handchirurgie, Universitätsklinikum Düsseldorf (Unknown)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, PD Dr. med. Christian Heiß, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15-035
Record Dates: First submitted 2017-06-22; First posted 2017-07-24 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Blue Light
Keywords: blue light; blood pressure; vascular function; endothelial function; health volunteers
MeSH Terms: interventions — Blue Light

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue light (Experimental): Each subject will be undergo a whole body exposure to blue light (453 nm wavelength) for 30 minutes.
  Interventions: Procedure: Blue light
- Control exposure (Placebo Comparator): Each participant will also undergo a control examination, where the body will be covered with a light tight foil during blue light exposure for 30 minutes.
  Interventions: Procedure: control exposure

INTERVENTIONS:
Procedure: Blue light — Subjects will be exposed to blue light (453 nm wavelength) for 30 minutes
  Arms: Blue light
Procedure: control exposure — Subjects will get control exposure to 30 minutes of whole body, which causes only comparable warming of skin as with blue light exposure.
  Arms: Control exposure

SUMMARY:
Ultraviolet light exposure was shown to be able to release nitric oxide from the skin into the blood stream and lead to an acute decrease in blood pressure and increase in vascular function. Additionally, preliminary work indicates that UV free blue light also releases nitric oxide in the skin mediating similar effects as seen with ultraviolet light A(UVA). It is the goal of the present experimental study to investigate the hemodynamic effects of whole body blue light exposure including blood pressure, endothelial function and vascular stiffness. Therefore, healthy volunteers will be exposed to 30 minutes whole body blue light (453 nm wavelength) and the change in blood pressure and endothelial function (Flow mediated dilation (FMD)), heart rate, forearm-blood flow, forearm vascular resistance central blood pressure and vascular stiffness ( pulse wave analysis by sphygmocor) will be measured.

In this randomized controlled cross-over study, 20 healthy subjects aged 30 to 60 years will participate.

ELIGIBILITY:
Inclusion Criteria:

* healthy, male subjects
* age between 30 and 60 years
* signed patient informed consent

Exclusion Criteria:

* diabetes mellitus
* acute inflammation (CRP >0.5mg/dl)
* cardiac arrythmia
* active cancer
* renal failure
* heart failure (NYHA II-IV)
* arterial hypotension (systolic pressure <100 mmHg)
* treatment with antihypertensive drugs
* dermatosis of the eyelid
* porphyria or hypersensitivity to porphyrins
* congenital or aсquired immune deficiency
* genetic conditions that cause an increased sensitivity to light or an increased risk to dermatological cancer (such as xeroderma pigmentosum, cockayne syndrome, bloom syndrome)
* previous intake or use of photosensitizing drugs, food or cosmetics (e.g. psychiatric medication, antibiotics, cardiovascular drugs, hormone, Hypericum, Bergamot orange) or use of perfumes

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change of peripheral blood pressure | baseline, during 30 min exposure and 2 hours thereafter
  Change of peripheral blood pressure as measured before, during and up to 2 hours after 30 min blue light as compared to control

SECONDARY OUTCOMES:
Change in endothelial function | baseline, during 30 min exposure and 2 hours thereafter
  measured by flow mediated dilation (FMD) before, immediately after 30 min exposure and at 2 h thereafter
Change from baseline heart rate | baseline, during 30 min exposure and 2 hours thereafter
  measured by electrocardiography (ECG) before, during and up to 2 hours after 30 min blue light as compared to control
Change from baseline forearm blood flow | baseline, during 30 min exposure and 2 hours thereafter
  measured by ultrasound before, immediately after 30 min exposure and at 2 h thereafter
Change from baseline forearm vascular resistance | baseline, during 30 min exposure and 2 hours thereafter
  measured by ultrasound before, immediately after 30 min exposure and at 2 h thereafter
Change from baseline central blood pressure | baseline, during 30 min exposure and 2 hours thereafter
  measured by applanation tonometry before, immediately after 30 min exposure and at 2 h thereafter
Change from baseline vascular stiffness | baseline, during 30 min exposure and 2 hours thereafter
  measured by applanation tonometry before, immediately after 30 min exposure and at 2 h thereafter
Change from baseline NO-species | baseline, during 30 min exposure and 2 hours thereafter
  determined by chemiluminescence before, immediately after 30 min exposure and at 2 h thereafter
Change from baseline Cortisol | baseline, during 30 min exposure and 2 hours thereafter
  measured before, immediately after 30 min exposure and at 2 h thereafter
Change from baseline Endorphins | baseline, during 30 min exposure and 2 hours thereafter
  measured before, immediately after 30 min exposure and at 2 h thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiß, MD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine, University Hospital Dusseldorf
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No